CLINICAL TRIAL: NCT02672397
Title: The Effect of a Culturally Sensitive Educational Intervention on Acceptance of Neuraxial Anesthesia in Hispanic and Caucasian Parturients: A Randomized Controlled Trial
Brief Title: The Effect of a Culturally Sensitive Educational Intervention on Acceptance of Neuraxial Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Brandon Togioka, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00010975
Record Dates: First submitted 2016-01-31; First posted 2016-02-03 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Labor Pain
Keywords: Epidural; Ethnicity; Education; Labor; obstetrical analgesia
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hispanic Intervention (Experimental): Hispanic subjects that receive additional epidural education [44 patients]
  Interventions: Behavioral: Additional Epidural Education
- Hispanic Control (No Intervention): Hispanic subjects that receive standard of care [44 patients]
- Non-Hispanic Intervention (Experimental): Non-Hispanic subjects that receive additional epidural education [44 patients]
  Interventions: Behavioral: Additional Epidural Education
- Non-Hispanic Control (No Intervention): Non-Hispanic subjects that receive standard of care [44 patients].

INTERVENTIONS:
Behavioral: Additional Epidural Education — All women allocated to receive additional epidural educational will be given a language appropriate pamphlet and video on neuraxial anesthesia. The video and pamphlet will be in the subject's primary language. After the subject watches the educational video they will be given an opportunity to go through the pamphlet with the research assistant and ask any questions they may have. For Spanish-speaking subjects this will occur through a telephone interpreter. The obstetric anesthesia providers and obstetricians caring for the subject will be absent for the educational video and post-video conversation.
  Arms: Hispanic Intervention; Non-Hispanic Intervention

SUMMARY:
The purpose of this study is to see if an educational intervention provided to pregnant women in early labor has an effect on their decision to use epidural anesthesia for relief of labor pain. The study will also investigate differences between Hispanic and non-Hispanic white women in their attitudes and beliefs regarding epidurals in labor. Previous studies have shown that Hispanic women receive epidural anesthesia in labor much less frequently than their non-Hispanic white counterparts. The investigators hypothesize that the rate of epidural use will be higher in subjects who receive the educational intervention than in those who do not.

Women who have been admitted to the OHSU labor and delivery unit will be screened for study eligibility. In order to minimize the influence of socioeconomic factors, only women receiving Medicaid will be enrolled. Other inclusion criteria include age of at least 18 years, having a fetus of at least 24 weeks gestational age, and being categorized as American Society of Anesthesiologist category 1 to 3. Exclusion criteria include any condition that either excludes or mandates neuraxial anesthesia. Midwife patients are also excluded from this study. Those who meet study criteria will be approached by a member of the study team and informed consent will be obtained.

Subjects will be randomly assigned to receive an educational intervention about epidurals or no educational intervention. Hispanic and non-Hispanic subjects will be randomized separately, yielding four study groups (Hispanic - intervention; Hispanic - control; non-Hispanic - intervention, non-Hispanic - control). The investigators expect to enroll approximately 176 women, 44 in each group.

All subjects will complete a survey in early labor and again 1 to 2 days postpartum that asks about common beliefs and misconceptions regarding epidurals. Subjects in the intervention group will receive an educational pamphlet and watch a video in their native language (spanish or english) about epidurals, and have an opportunity to ask questions. Study staff will collect limited information about the subject's labor and delivery from the electronic medical record.

DETAILED DESCRIPTION:
Study Design

This study is designed to be a prospective, single-blinded, randomized controlled trial at Oregon Health and Science University (OHSU) in Portland, Oregon. The investigators will enroll Hispanic and non-Hispanic parturients in equal numbers on the labor and delivery floor to receive both an educational pamphlet and video in their primary language or no educational intervention. All parturients will receive standard of practice consent for general/regional anesthesia by an anesthesiology resident or attending.

Study Population

A total of 176 participants will be enrolled in the study. Within the 176 participants there will be four groups of patients: (1) Hispanic subjects that receive additional epidural education [44 patients], (2) Hispanic subjects that receive standard of care [44 patients], (3) non-Hispanic subjects that receive additional epidural education [44 patients], and (4) non-Hispanic subjects that receive standard of care [44 patients].

Over the past year 421 Hispanic and 215 non-Hispanic patients with Medicaid insurance delivered at OHSU. The rate-limiting step in the study will be enrolling enough non-Hispanic subjects on Medicaid and so study timeline calculations are based upon expected enrollment of those subjects. Assuming 15% of patients approached decline study participation and the research team misses another 35% of patients the investigators believe they can enroll the necessary 88 subjects in 300 days or approximately 10 months (during which time 177 non-Hispanic Medicaid deliveries would occur).

Patients appropriate for inclusion in the study will be identified at OHSU after they have been admitted to the labor and delivery unit. A cursory review of the labor and delivery unit census on EPIC will be used to identify qualifying patients (ASA I-III category patients of 18 years of age on Medicaid with that are either in labor or committed to labor via induction). All patients who pass this initial screen with have a more thorough review of their record with particular attention paid to ethnicity and medical conditions that would affect the decision to offer neuraxial analgesia.

Setting

Informed consent, Initial Encounter survey, and Epidural Pre-Test Questionnaire will be administered in the OHSU Labor and Delivery Unit. The Epidural Post-Test Questionnaire will be administered in the patient's recovery room 1-2 days after giving birth.

Recruitment Methods

Patients that appear to meet inclusion criteria will be identified at OHSU after they have been admitted to the labor and delivery unit. A cursory review of EPIC on the work computers of the researchers or labor and delivery unit computers will be used to identify patients that warrant a deeper chart review (ASA I-III category patients of at least 18 years on Medicaid that are either in labor or committed to labor via induction). All patients that pass this initial screen will have a more thorough review of their medical record with particular attention paid to ethnicity, whether they are an MD or midwife patient, and medical conditions that may affect the decision to offer neuraxial anesthesia. All patients that pass this EPIC screen will be approached by the research team and allowed to participate in the study. There will be no fliers, advertisements, videos, or webpages set up to recruit patients. There will be no monetary awards or free services offered to study participants.

Consent Process

A member of the research team will perform subject recruitment and obtain written informed consent in the OHSU Labor and Delivery Unit in order to minimize the possibility of coercion.

Patients will be provided the Consent and Authorization form in their preferred language (English or Spanish) and will have an opportunity to ask questions of the research team member after the study protocol is explained. An interpreter/translator will be available via telephone for Spanish speaking women during this time.

Procedures

Subject allocation will occur in the labor room after informed consent has occurred. Allocation will occur when the research assistant opens one of a series of sequentially numbered opaque envelopes containing group assignment (by a computer generated random number sequence [Excel, Redmond WA]. A researcher not involved in either subject enrollment or subject assignment will generate the random number sequence. The anesthesia and obstetric team caring for the subject will remain blinded on whether the subject received additional educational materials; however, due to the type of study it is impossible to blind the subject. Subjects will be allocated to either an epidural-focused educational intervention or no intervention by ethnicity stratified block randomization.

Subjects that agree to participate in the study will have demographic data collected from EPIC (age, race, gravida, parity, gestational age, BMI, birth history) and will be given a subject questionnaire in their primary language that will ask about potential confounders that may affect epidural usage (highest education achieved, length of time the subject's family has lived in the U.S., past personal and family experience with epidurals, needle phobia, etc.). At the conclusion of the study some additional information will be taken from EPIC (length of labor, type of delivery, APGAR scores, and whether an epidural was used for labor analgesia).

All subjects enrolled in the study will be given a survey in their primary language seeking to identify potential barriers to neuraxial anesthesia utilization. Included in this survey will be a yes/no checklist for the subject to complete that includes some previously published reasons that patients commonly give for not wanting neuraxial anesthesia. This survey will be given again in the postpartum period to all women enrolled in the study. The postpartum survey will serve as a post-test to evaluate the effectiveness of the educational intervention in those women that received additional education materials. The post-test will also be given to women in the control group to determine if the process of delivering a baby either with or without an epidural affects subject views on neuraxial anesthesia. The completion of the posttest will mark the end of each parturient's time of participation in the study.

All women allocated to receive additional educational materials will be given a language appropriate pamphlet and video on neuraxial anesthesia. The video and pamphlet will be in the subject's primary language. After the subject watches the educational video they will be given an opportunity to go through the pamphlet with the research assistant and ask any questions they may have. For Spanish-speaking subjects this will occur through a telephone interpreter. The obstetric anesthesia providers and obstetricians caring for the subject will be absent for the educational video and post-video conversation.

Women who elect to receive neuraxial anesthesia will be administered the procedure by an anesthesiology resident with supervision by an attending anesthesiologist. A lumbar epidural catheter will be placed and after initial bolus (spinal or epidural) all subjects will be started on a patient-controlled epidural analgesia (PCEA) protocol with a solution of 0.055% bupivacaine with 1 mcg/mL sufentanil. The initial PCEA settings for all subjects will be the following: maintenance infusion rate of 10 ml/hr, bolus of 5 ml, lockout of 15 minutes, with a maximum of 4 boluses an hour. The maintenance infusion rate, bolus volume, and lockout interval will be allowed to be adjusted as deemed necessary by the obstetric anesthesiology team. Subjects with pain refractory to the initial PCEA settings will be allowed to get additional epidural boluses of medication by the anesthesiology resident or attending. The PCEA will be continued until delivery or slightly thereafter depending upon subject need. The PCEA will be allowed to be turned off or down to help with stage two pushing or to avoid maternal hypotension. Other more rare complications involving neuraxial anesthesia will be dealt with according to standard of care practice.

Data Analysis

Sample size calculations are based upon the abstract presented at the Society for Maternal-Fetal Medicine. In that study, only 40% of women assigned to additional prenatal epidural education classes attended the prescribed intervention. With 40% attendance the authors of the study found a 14% difference in epidural utilization rates. Subjects in this study will be randomized on labor and delivery after hospital admission. The investigators estimate that 90% of women will get the assigned educational intervention. Assuming epidural education has the same effect in this study as that seen in the abstract by Kanter et al. the investigators expect to see a 31% increase in epidural utilization. Based upon data at OHSU from June 2013 to May 2014 the current epidural rate at OHSU for Hispanics is 45.3% and the current epidural rate for non-Hispanics is 55.8%. Assuming a 31% difference in epidural usage in the Hispanic population after implementation of the study protocol, with an alpha of 0.05 and a power of 80%, 44 subjects would need to be randomized to each of four groups.

The investigators will compare the intervention to control group within both the Hispanic and non-Hispanic populations on the primary outcome of neuraxial anesthesia utilization using the chi-squared statistic. Pre and post delivery scores from the Neuraxial Anesthesia Survey will be compared using the Wilcoxon signed-rank test. Subject characteristics between study arms will be compared to one another with the chi-squared statistic or Fisher's Exact Test for categorical outcomes and the student t test, or a non-parametric equivalent, for continuous variables. A p < 0.05 will be required to reject the null hypothesis that no difference between epidural utilization rates exists between those that received the educational intervention and those that did not.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Pregnant with a fetus > 24 weeks gestation
* Medicaid insurance
* ASA class 1 to 3
* Arriving at OHSU in spontaneous labor, requiring induction, or receiving augmentation of labor

Exclusion Criteria:

* Patients having scheduled cesarean sections
* Patients with conditions that are contraindications for epidural labor analgesia
* Patients in whom epidural analgesia is mandated by the medical team
* Patients delivering with a midwife

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2017-02-25 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Epidural usage rate | 1 year
  The primary aim of this study is to determine if women that receive focused education on epidural labor pain management in the form of a pamphlet and video are more likely to decide to use an epidural. The investigators will also compare the effect of the intervention on hispanic women to the effect of the intervention on non-hispanic women.

SECONDARY OUTCOMES:
Pre and post intervention Beliefs about Epidurals Questionnaire | 1 year
  A secondary goal of this study is to determine if the intervention changes women's beliefs about epidural labor pain management

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M Togioka, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU Labor and Delivery; Oregon Health and Science University Hospital, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rust G, Nembhard WN, Nichols M, Omole F, Minor P, Barosso G, Mayberry R. Racial and ethnic disparities in the provision of epidural analgesia to Georgia Medicaid beneficiaries during labor and delivery. Am J Obstet Gynecol. 2004 Aug;191(2):456-62. doi: 10.1016/j.ajog.2004.03.005. PMID 15343221
- [Background] Glance LG, Wissler R, Glantz C, Osler TM, Mukamel DB, Dick AW. Racial differences in the use of epidural analgesia for labor. Anesthesiology. 2007 Jan;106(1):19-25; discussion 6-8. doi: 10.1097/00000542-200701000-00008. PMID 17197841
- [Background] Toledo P, Sun J, Grobman WA, Wong CA, Feinglass J, Hasnain-Wynia R. Racial and ethnic disparities in neuraxial labor analgesia. Anesth Analg. 2012 Jan;114(1):172-8. doi: 10.1213/ANE.0b013e318239dc7c. Epub 2011 Nov 10. PMID 22075013